CLINICAL TRIAL: NCT03547453
Title: Ovarian Ultrasonography for the Clinical Evaluation of Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Cornell University (Other)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: 00070269
Record Dates: First submitted 2018-05-09; First posted 2018-06-06 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Polycystic Ovary Syndrome (PCOS); Menstrual Irregularity; Overweight and Obesity
Keywords: Menstrual cycles; Ultrasound; Ovary; Polycystic Ovary Syndrome (PCOS)
MeSH Terms: conditions — Polycystic Ovary Syndrome; Menstruation Disturbances; Overweight; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum samples not containing DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Regular Menstrual Cycles: Women will be assigned to this category if they report a history of regular menstrual cycles (every 21 to 35 days). Recruitment will be targeted to obtain 20 lean (BMI<25 kg/m2) and 20 overweight or obese (BMI>24.9kg/m2) women in each of the following age groups: 18-24y (early), 25-34y (mid), ≥35y (later adulthood).
- Polycystic Ovarian Syndrome: Women will be assigned to this category if they have clinical or biochemical androgen excess and report a history of irregular menstrual cycles (<21 days or >35 days), including women with a pre-existing diagnosis of PCOS. Recruitment will be targeted to obtain 20 lean (BMI<25kg/m2) and 20 overweight or obese (BMI>24.9kg/m2) women in each of the following age groups: 18-24y (early), 25-34y (mid), ≥35y (later adulthood).

SUMMARY:
The investigators would like to determine how aspects of adiposity and age influence ultrasound features of the ovaries which are used to diagnose polycystic ovarian syndrome (PCOS). The study will also compare anti-Müllerian hormone (AMH) levels against ultrasound features of the ovary to predict PCOS.

DETAILED DESCRIPTION:
The purpose of this study is to develop ultrasound criteria for polycystic ovaries for women with PCOS across early, mid and late adulthood and to assess the impact of body composition on these ultrasound criteria.. The study will also compare ultrasound features of the ovary against or in combination with AMH (a hormonal biomarker) in predicting PCOS. This research will help improve the diagnosis of PCOS by considering multiple markers (i.e., ultrasound features and AMH levels) and multiple modifiers of those markers (i.e., age and adiposity).

As the name implies, the primary ultrasound feature used to diagnose PCOS is polycystic ovaries (PCO). However, PCO have frequently been observed in healthy women, calling into question the specificity of PCO to the condition of PCOS, as well as its ability to inform progression of the disease and/or response to treatment. The Lujan laboratory recently showed that the most widely accepted ultrasound criteria for PCO overlap with features of the normal ovary, and their laboratory proposed new thresholds to redefine PCO. These new criteria represented a significant change in the definition of PCO owing to the improved resolution of new technology. That said, these new criteria are still limited. They do not account for factors known or suspected to influence ovarian morphology. For example, follicle counts and ovarian size increase at puberty and decrease with age. Additional results from the Lujan laboratory showed that follicle number per ovary (FNPO) thresholds for women in later adulthood (35-38y) were substantially lower than those in early (18-25y) and mid-adulthood (26-34y). Furthermore, the new criteria for PCO do not account for a potential impact of adiposity on ovarian morphology. In the same study, conducted by the Lujan laboratory, overweight women exhibited more 6-9mm follicles than lean women, irrespective of androgen status.

Lastly, there is significant interest in determining whether AMH can serve as a surrogate to sonographic measures to define PCO. AMH is a peptide hormone produced by the granulosa cells of growing follicles and circulating levels represent secretions by antral follicles ≤8mm. Accordingly, serum AMH is increased in women with PCOS, reflecting the accumulation of 2-5mm antral follicles and greater production by granulosa cells of PCO compared to normal ovaries. Excess AMH is thought to inhibit follicle growth and selection. Unlike discrete aspects of ovarian morphology (i.e. follicle number or size),85 AMH levels remain largely constant throughout the normal menstrual cycle.Such stability may make AMH a more advantageous functional and surrogate morphological indicator of ovarian status compared to morphologic features. Further, some have argued that the variability in ultrasound assessments, and unsuitability of transvaginal approaches in certain clinical populations, justify the pursuit of a less onerous biomarker of PCO. However, there is significant bias across AMH assays and a consensual threshold for AMH to define PCO has not been determined. Proposed thresholds were hindered by heterogeneity in assay performance and in the clinical cohorts assessed. Ultimately, the ability of AMH to serve as a surrogate marker for PCO remains unknown and should be evaluated against sonographic measures in well-defined cohorts with improved assays. In this study, the researchers plan to refine the sonographic definition of PCO by establishing age-specific criteria that maintain sensitivity and specificity for PCOS in both lean and overweight populations. They will also clarify any ability of anti-Müllerian hormone (AMH) to better inform the diagnosis of PCOS.

To accomplish these objectives, the investigators plan to recruit 120 women with regular ovulatory cycles and 120 women with PCOS. Within each of these categories, the investigators plan to recruit 20 lean and 20 overweight women in each age group: 18-24y (early), 25-34y (mid), ≥35y (later adulthood). Ultrasound scans of the ovaries will be assessed for the total number, size, and distribution of follicles using both two- and three-dimensional imaging techniques. Additionally, participants will have blood samples collected to determine serum concentrations of AMH. Because features of the ovaries are expected to be different in lean and overweight women, the researchers hope to develop ultrasound criteria that will help healthcare providers to diagnosis specific ovulation problems in women across all body sizes and ages. This project addresses the need to improve methods and criteria used to define PCO across clinical populations.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years
* At least 2y post-menarche
* BMI >18.5kg/m2
* Good visibility of the ovaries on ultrasound
* Pelvic exam with normal results within the last 2 years

Either:

* Regular menstrual cycles (21-35 days);
* Irregular menstrual cycles (>36 days); or
* Previous diagnosis of PCOS from a primary care provider

Exclusion Criteria:

* Use of medication(s) known or suspected to interfere with reproductive function, metabolism, and/or appetite (e.g., oral contraceptives) within the past 3 months
* Use of fertility medications in the past 2 months (e.g., Clomid)
* Current use of a non-copper intrauterine device for contraception (e.g., Mirena)
* Diagnosis of premature ovarian failure, endometriosis, or another disease/disorder (other than PCOS) known or suspected to interfere with reproductive function
* History of ovarian surgery
* Missing uterus or an ovary
* Pregnant or breastfeeding
* Diagnosis of a bleeding disorder
* Regular use of blood thinners/anticoagulants
* Skin allergy/condition that might be aggravated by alcohol application
* Currently being treated for a vaginal infection, cervical infection, sexually transmitted infection, or disease either with antibiotics, antifungals, or anti-viral medication
* Abnormal vaginal discharge, pelvic pain, and/or blisters/lesions/warts/skin growths in the genital/anal area, which have not been examined by a medical professional.
* Vaginal abnormality (e.g., vaginal atresia/hypoplasia, vaginal septation, Mullerian agenesis, vulvar/vaginal malignancy).
* Not otherwise healthy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women must be able to transport to the University of Rochester. Eligible participants are older than 18 years with a BMI of 18.5 kg/m2 or higher. Women are screened and enrolled following consent based on their response to our advertisements. Enrollment is restricted to the geographical area.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Follicle number per ovary | 1 day
  The number of follicles in each ovary will be assessed by ultrasonography

SECONDARY OUTCOMES:
Follicle number per cross section | 1 day
  The number all follicles in a single cross sectional plane of each ovary will be assessed by ultrasonography
Ovarian volume | 1 day
  The size of each ovary will be determined by ultrasonography for each participant and compared across groups.
Stromal echogenicity on ultrasound | 1 day
  The brightness of the ovarian stroma in a single cross section will be determined by ultrasonography for each participant and compared across groups.
Ovarian area-stromal area ratio | 1 day
  The ratio of the stromal area to the total ovarian area of the ovary in a single cross section will be determined by ultrasonography for each participant and compared across groups.
Follicle distribution pattern | 1 day
  The follicle distribution pattern will be assessed by ultrasonography for each participant and compared across groups.
Anti-Müllerian hormone | 1 day
  Circulating AMH levels in the serum will be determined for each participant and compared across groups.
LH-FSH ratio | 1 day
  The ratio of circulating LH to FSH concentrations in the serum will be determined for each participant and compared across groups
Hirsutism Score | 1 day
  Degree of hirsutism as judged by the Ferriman-Gallwey scale will be determined and compared across groups
Androgen concentrations | 1 day
  Total testosterone, androstenedione and free androgen index concentrations in serum will be determined and compared across groups.
Menstrual Cycle Length | 1 day
  Average menstrual cycle length as determined by self-reported history will be determined and compared across groups
Body mass index | 1 day
  The ratio of weight to height will be determined and compared across groups.
Waist-to-hip ratio | 1 day
  The ratio of waist circumference to hip circumference will be determined and compared across groups.

CONTACTS AND LOCATIONS:
Overall Officials: Marla E. Lujan, PhD, Principal Investigator — Cornell University; Kathleen Hoeger, MD, Principal Investigator — University of Rochester
Locations (1):
- Strong Fertility Center, Rochester, New York, United States